CLINICAL TRIAL: NCT03550144
Title: Effects of Awe on Mental Health and Well-Being
Brief Title: Improving Mental Health and Well-Being Via Awe Walks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-20001
Record Dates: First submitted 2018-05-16; First posted 2018-06-08 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Awe; Compassion; Anxiety
Keywords: Awe; Compassion; Anxiety; Positive emotions; Aging
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awe Walk Condition (Experimental): Participants were instructed to take at least one (~15 minute) walk per week for 8 consecutive weeks. Participants were told to seek the experience of feeling awe. Participants were told to keep a fairly light to moderate pace and were encouraged to walk alone and without interruption from a mobile device.
  Interventions: Behavioral: Awe Walk
- Control Walk Condition (Active Comparator): Participants were instructed to take at least one (~15 minute) walk per week for 8 consecutive weeks. Participants were told to keep a fairly light to moderate pace and were encouraged to walk alone and without interruption from a mobile device.
  Interventions: Behavioral: Control Walk

INTERVENTIONS:
Behavioral: Awe Walk — To examine the effect of weekly awe walks in cognitively healthy older adults.
  Arms: Awe Walk Condition
Behavioral: Control Walk — To examine the effect of weekly walks in cognitively healthy older adults.
  Arms: Control Walk Condition

SUMMARY:
Awe is a powerful positive emotion that offsets negative emotion and fosters prosocial behavior. This study examined the effects of awe on health and well-being in healthy older adults. Half of the participants took a weekly "awe walk" while the other half took a weekly walk with no further instructions.

DETAILED DESCRIPTION:
Awe fosters well-being and positive emotions that promote social relationships. Awe shifts attention from ourselves to the outside world and is associated with diminished self-focused attention. We aimed to increase awe in healthy older adults to test whether greater awe experience would lead to gains in other types of positive emotional experience and reductions in negative emotional experience.

ELIGIBILITY:
Inclusion Criteria:

* Stable medical condition for 3 months prior to screening
* Reliant informant with frequent contact with participant who is available to provide observations of participant
* Fluent in English or Spanish
* Age: 40 and above
* Able to complete baseline assessments
* Education or work history sufficient to exclude mental retardation
* Physically acceptable for this study as confirmed by medical history, physical exam, neurological exam and clinical tests

Exclusion Criteria:

* Major memory concerns/diagnosed memory condition
* Korsakoff encephalopathy
* Active substance abuse
* Brain tumor
* Active neoplastic disease (skin tumors other than melanoma are not exclusionary)
* Parkinson's disease
* Multiple sclerosis (untreated)
* Sleep apnea
* History of clinically significant stroke
* Current evidence or history in the past 2 years of epilepsy, focal brain lesion, cancer, steroid use, or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
* Blindness, deafness, language difficulties or any other disability which may prevent the participant from participating or cooperating in the protocol

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2018-05-26 (Actual)

PRIMARY OUTCOMES:
Daily awe experience questionnaire | 8 weeks
  Increase in awe experience

SECONDARY OUTCOMES:
Daily compassion experience questionnaire | 8 weeks
  Increase in daily compassion experience
Daily negative emotional experience questionnaire | 8 weeks
  Decrease in daily negative emotional experience
Generalized Anxiety Disorder- 7 Item Scale | 8 weeks
  Decrease in anxiety
Satisfaction With Life Scale | 8 weeks
  Increase in well-being

CONTACTS AND LOCATIONS:
Overall Officials: Virginia E Sturm, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Memory and Aging Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Keltner D, Haidt J. Approaching awe, a moral, spiritual, and aesthetic emotion. Cogn Emot. 2003 Mar;17(2):297-314. doi: 10.1080/02699930302297. PMID 29715721
- [Background] Kaup AR, Byers AL, Falvey C, Simonsick EM, Satterfield S, Ayonayon HN, Smagula SF, Rubin SM, Yaffe K. Trajectories of Depressive Symptoms in Older Adults and Risk of Dementia. JAMA Psychiatry. 2016 May 1;73(5):525-31. doi: 10.1001/jamapsychiatry.2016.0004. PMID 26982217
- [Background] Williams JE, Paton CC, Siegler IC, Eigenbrodt ML, Nieto FJ, Tyroler HA. Anger proneness predicts coronary heart disease risk: prospective analysis from the atherosclerosis risk in communities (ARIC) study. Circulation. 2000 May 2;101(17):2034-9. doi: 10.1161/01.cir.101.17.2034. PMID 10790343
- [Background] Fredrickson BL, Cohn MA, Coffey KA, Pek J, Finkel SM. Open hearts build lives: positive emotions, induced through loving-kindness meditation, build consequential personal resources. J Pers Soc Psychol. 2008 Nov;95(5):1045-1062. doi: 10.1037/a0013262. PMID 18954193
- [Background] Stellar JE, John-Henderson N, Anderson CL, Gordon AM, McNeil GD, Keltner D. Positive affect and markers of inflammation: discrete positive emotions predict lower levels of inflammatory cytokines. Emotion. 2015 Apr;15(2):129-33. doi: 10.1037/emo0000033. Epub 2015 Jan 19. PMID 25603133
- [Background] Diener E, Chan MY. Happy people live longer: Subjective well-being contributes to health and longevity. .Applied Psychology: Health and Well-Being 2011;3:1-43
- [Background] Levenson RW, Ascher E, Goodkind M, McCarthy M, Sturm V, Werner K. Chapter 25 Laboratory testing of emotion and frontal cortex. Handb Clin Neurol. 2008;88:489-98. doi: 10.1016/S0072-9752(07)88025-0. No abstract available. PMID 18631708
- [Background] Emmons RA, McCullough ME. Counting blessings versus burdens: an experimental investigation of gratitude and subjective well-being in daily life. J Pers Soc Psychol. 2003 Feb;84(2):377-89. doi: 10.1037//0022-3514.84.2.377. PMID 12585811
- See also: Greater Good Science Center — https://greatergood.berkeley.edu/
- See also: Global Brain Health Institute — http://www.gbhi.org/

DOCUMENTS (2):
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03550144/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03550144/SAP_001.pdf